CLINICAL TRIAL: NCT05406141
Title: Nutrition Sufficiency, Allergy Efficacy and Safety of an Amino Acid-Based Formula Neocate Jr in Children With Food Protein Allergy
Brief Title: Nutrition Sufficiency, Allergy Efficacy and Safety of Neocate Jr in Children With Food Protein Allergy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Children's Hospital (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202107 V2.0
Record Dates: First submitted 2022-03-14; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-02

CONDITIONS: Food Allergy in Children; Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children with food protein allergy (Experimental)
  Interventions: Dietary Supplement: Amino acid formula (Neocate Jr)

INTERVENTIONS:
Dietary Supplement: Amino acid formula (Neocate Jr) — Use Neocate Jr for 4 weeks, either as sole source of nutrition or oral nutritional supplement:
  * Sole source of nutrition: as far as possible >7 days, especially newly diagnosed allergy children
  * Oral nutritional supplement (Neocate Jr ≥50% of daily total energy and the rest provided by food)

SUMMARY:
The main purpose of this study is to evaluate efficacy and safety of an amino acid-based formula Neocate Jr in children with food protein allergy, and to evaluate nutrition sufficiency of Neocate Jr in 1 to 10 years old children with food protein allergy.

DETAILED DESCRIPTION:
This is an open, self-controlled multi-center clinical study. Target population is 1～10 years old children allergic to cow's milk and/or food protein, confirmed by pediatrician. The study plans to recruit about 50 subjects to have an intervention period of 4 weeks. Data will be collected at baseline, week 1, 2 and 4. The hypothesis is that the amino acid formula (Neocate Jr) is effective in relieving food protein allergy symptoms, and meanwhile supporting normal growth in children with food protein allergy. Efficacy parameters are the the improvement of food protein allergy symptoms (SCORAD score, serum IgE), growth and development index (weight, height, weight for height), and nutrition related labs (such as hemoglobin, total blood protein, albumin, pre-albumin).

ELIGIBILITY:
Inclusion Criteria:

* 1～10 years old
* The children with cow's milk/food protein allergy confirmed by pediatrician including sequential feeding/newly diagnosed children, and children with Eosinophilic Esophagitis, Gastroesophageal reflux disease, Food Protein-Induced Enterocolitis Syndrome (clinical symptoms and signs, IgE, oral food challenge, etc.)
* Stable Vital Signs
* Written informed consent from the children's parents/guardian

Exclusion Criteria:

* Allergic to any ingredient in the recipe
* GI function failure
* Complete obstruction of the digestive tract
* Intractable diarrhea
* Noncooperation of neurologic or mental diseases
* Disapproval of pediatricians

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
SCORAD score | Change from baseline SCORAD score to Neocate Jr feeding at day 28
  SCORing Atopic Dermatitis (SCORAD) evaluation scale is selected as the indicator of allergy symptoms improvement, and will be evaluated by the investigator at each visit. The SCORAD score range is between 0 and 103, and lower scores mean a better outcome.
serum IgE | Change from baseline serum IgE to Neocate Jr feeding at day 28
  Serum IgE is selected as an indicator of allergy improvement, and will be measured by the investigator at baseline and day 28 for comparison.
weight for age | Change from baseline body weight to Neocate Jr feeding at day 28
  Body weight for age is selected as the primary indicator of nutrition sufficiency, and will be measured by the investigator at each visit, and compared to World Health Organization (WHO) standard.

SECONDARY OUTCOMES:
weight for height | Change from baseline to Neocate Jr feeding at day 28
  Weight for height is selected as the an indicator of nutrition sufficiency, and will be evaluated by the investigator at each visit.
hemoglobin, total blood protein, albumin, pre-albumin | Change from baseline to Neocate Jr feeding at day 28
  Hemoglobin, total blood protein, albumin and pre-albumin are selected as indicators of nutrition sufficiency, and will be measured by the investigator at baseline and day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Zailing Li, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China